CLINICAL TRIAL: NCT03268122
Title: Comparison of Standard Isolation With Targeted Isolation for Preventing Nosocomial Transmission of MRSA and VRE: A Pilot Clinical Trial
Brief Title: Comparison of Standard Isolation With Targeted Isolation for Preventing Nosocomial Transmission of MRSA and VRE
Acronym: CONTACT-PILOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Todd Rice, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 161137
Record Dates: First submitted 2017-08-09; First posted 2017-08-31 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: MRSA; VRE Infection
Keywords: Patient Isolation; Methicillin-Resistant Staphylococcus aureus; Vancomycin-Resistant Enterococci

STUDY DESIGN:
Intervention Model Description: Multiple-crossover, cluster-randomized, controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Contact Isolation (Active Comparator): Patients in the standard contact isolation arm will be under the standard contact isolation strategy during the entire time they are physically located in the Medical ICU.
  Interventions: Other: Standard Contact Isolation
- Targeted Contact Isolation (Active Comparator): Patients in the targeted contact isolation arm will be under the targeted contact isolation strategy during the entire time they are physically located in the Medical ICU.
  Interventions: Other: Targeted Contact Isolation

INTERVENTIONS:
Other: Standard Contact Isolation — With regards to MRSA and VRE, the wearing of gowns and gloves will be required for all staff entering a patient room if the patent has an infection or colonization with MRSA or VRE or a recent history (within 90 days) of either
  Other Names: Standard Contact Precautions
  Arms: Standard Contact Isolation
Other: Targeted Contact Isolation — With regards to MRSA and VRE, the wearing of gowns and gloves will be required for all staff entering a patient room if the patient has an active, highly-transmissible infection with MRSA and/or VRE.
  A highly-transmissible infection is defined as one with uncontained secretions or excretions (diarrhea, vomiting, or open draining wounds) or pneumonia.
  Other Names: Targeted Contact Precautions
  Arms: Targeted Contact Isolation

SUMMARY:
Hospital-acquired infections are common and frequently lead to poor outcomes, including death, in affected patients. Two common organisms that cause infections in the hospital are methicillin-resistant Staphylococcus aureus (MRSA) and vancomycin-resistant Enterococcus (VRE). One strategy used to prevent these infections is contact isolation of hospitalized patients with MRSA and/or VRE. It is unclear whether contact isolation decreases the rate of infection with MRSA and/or VRE. The CONTACT-PILOT study is designed to test the hypothesis that contact isolation decreases the rate of infection with MRSA and/or VRE in patients in the intensive care unit (ICU). The study will enroll all adults in the Medical ICU and will run between September 2017 and April 2018. During some months, all patients in the Medical ICU patients will be placed in isolation for MRSA or VRE if they have a current infection or colonization with either organism, or a recent history thereof. During other months, patients will only be placed in isolation for MRSA or VRE if they have an active, highly-transmissible infection with either organism, such as a pneumonia or an open, draining wound.

DETAILED DESCRIPTION:
CONTACT-PILOT is a single center, pilot, multiple crossover, cluster-randomized trial of contact isolation for MRSA and VRE in the Vanderbilt Medical Intensive Care Unit (MICU) in order to determine if contact isolation reduces the rate of ICU-acquired infection with MRSA and/or VRE. Specifically, the study will randomly assign the entire MICU to one of two contact isolation strategies for 2 months, and then switch the entire MICU over to the second strategy. The first strategy is the current practice, also referred to as standard contact isolation, which is to place all patients with MRSA and/or VRE infection or colonization (or a history of either) on contact isolation. The second strategy is targeted contact isolation, in which patients with MRSA and/or VRE would only be placed on contact isolation if they have an active infection with one (or both) of these organisms with a high risk of transmission, such as an open, draining wound or a pneumonia. The study will be divided into four alternating 2-month treatment blocks, two for each strategy, with one "run-in" week at the start of each treatment block in order to transition between the two treatment strategies, for a total study duration of 8 months. The interventions will occur between September 1, 2017 and April 30, 2018. All adult MICU patients will be enrolled in the study. The primary outcome will be the rate of new ICU-acquired MRSA and VRE infections. Data analysis will be performed using a pre-specified data analysis plan. This study is being performed as a preliminary study to evaluate the feasibility and safety of the study plan.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the study ICU, the Vanderbilt University Medical Center Medical Intensive Care Unit, during an active enrollment period

Exclusion Criteria:

* Age less than 18 years old
* Patients admitted during a run-in period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1974 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Composite rate of ICU-acquired MRSA or VRE infections | 48 hours after enrollment to 48 hours after study ICU discharge, censored at 28 days after enrollment
  The primary endpoint is defined as an MRSA or VRE infection in a patient not currently diagnosed with or being treated for that infection at least 48 hours after admission to the study ICU and while the patient either remains in the study ICU or is within 48 hours of discharge or transfer from the study ICU, truncated at day 28 after enrollment. The composite rate will be reported in infections per 1000 patient-days.

SECONDARY OUTCOMES:
Rate of ICU-acquired MRSA infection | 48 hours after enrollment to 48 hours after study ICU discharge, censored at 28 days after enrollment
  An MRSA infection in a patient not currently diagnosed with or being treated for that infection at least 48 hours after admission to the study ICU and while the patient either remains in the study ICU or is within 48 hours of discharge or transfer from the study ICU, truncated at day 28 after enrollment. The rate will be reported in infections per 1000 patient-days.
Rate of ICU-acquired VRE infection | 48 hours after enrollment to 48 hours after study ICU discharge, censored at 28 days after enrollment
  A VRE infection in a patient not currently diagnosed with or being treated for that infection at least 48 hours after admission to the study ICU and while the patient either remains in the study ICU or is within 48 hours of discharge or transfer from the study ICU, truncated at day 28 after enrollment. The rate will be reported in infections per 1000 patient-days.
Rate of ICU-acquired MRSA bacteremia | 48 hours after enrollment to 48 hours after study ICU discharge, censored at 28 days after enrollment
  A positive clinical blood culture for MRSA in a patient not currently diagnosed with or being treated with that infection at least 48 hours after admission to the study ICU and while the patient either remains in the study ICU or is within 48 hours of discharge or transfer from the study ICU, truncated at day 28 after enrollment. The rate will be reported in infections per 1000 patient-days.
Rate of ICU-acquired VRE bacteremia | 48 hours after enrollment to 48 hours after study ICU discharge, censored at 28 days after enrollment
  A positive clinical blood culture for VRE in a patient not currently diagnosed with or being treated for that infection at least 48 hours after admission to the study ICU and while the patient either remains in the study ICU or is within 48 hours of discharge or transfer from the study ICU, truncated at day 28 after enrollment. The rate will be reported in infections per 1000 patient-days.
Composite rate of ICU-acquired MRSA or VRE bacteremia | 48 hours after enrollment to 48 hours after study ICU discharge, censored at 28 days after enrollment
  A clinical blood culture positive for either MRSA or VRE in a patient not currently diagnosed with or being treated for that infection at least 48 hours after admission to the study ICU and while the patient either remains in the study ICU or is within 48 hours of discharge or transfer from the study ICU, truncated at day 28 after enrollment. The composite rate will be reported in infections per 1000 patient-days.
Composite rate of hospital-acquired MRSA or VRE infection | 48 hours after enrollment to 48 hours after study hospital discharge, truncated at 28 days after enrollment
  An MRSA or VRE infection in a patient not currently diagnosed with or being treated for that infection at least 48 hours after admission to the study ICU and while the patient either remains admitted to the study hospital or is within 48 hours of discharge or transfer from the study hospital, truncated at day 28 after enrollment. The composite rate will be reported in infections per 1000 patient-days.
Composite rate of hospital-acquired CLABSI, CAUTI, BSI, Clostridium difficile infection, and VAP. | 48 hours after enrollment to 48 hours after study ICU discharge, truncated at day 28 after enrollment (except for Clostridium difficile infections, which are truncated at the time of study ICU discharge)
  Composite rate of certain healthcare-associated infections: central line-associated bloodstream infection (CLABSI), catheter-associated urinary tract infection (CAUTI), bloodstream infection (BSI), Clostridium difficile infection, and ventilator-associated pneumonia (VAP) in patients not currently diagnosed with or being treated for those infections, truncated at day 28 after enrollment.
28-day mortality | Date of enrollment until 28 days after enrollment
  All-cause mortality up until 28 days after enrollment, censored at hospital discharge
In-hospital mortality | Date of enrollment until hospital discharge, censored at 28 days after enrollment
  All-cause death while admitted to the study hospital, truncated 28 days after enrollment
ICU mortality | Date of enrollment until study ICU discharge, censored at 28 days after enrollment
  All-cause death while admitted to the study ICU, truncated 28 days after enrollment
ICU length of stay | Study enrollment until study ICU discharge, truncated at 28 days after enrollment
  Length of Stay in the ICU
Hospital length of stay | Study enrollment until study hospital discharge, truncated at 28 days after enrollment
  Length of Stay in the Hospital
Proportion compliant with hand hygiene | Up to 8 months
  Compliance by staff members with hand hygiene will be defined as using alcohol-based foam and/or soap and water immediately before entering a patient room and immediately after exiting a patient room, unless the patient specifically requires soap and water to be utilized after exiting their patient room (e.g. a patient with Clostridium difficile infection), in which case compliance after exiting that patient room would only be achieved by handwashing with soap and water.
Proportion compliant with contact isolation | Up to 8 months
  Compliance with contact isolation precautions by staff members will be defined as donning gown and gloves immediately prior to entering a patient room and removal of both of these items immediately before exiting a patient room.
Estimated cost of gowns and gloves | Up to 8 months
  This outcome will be calculated from the rate of gowns and gloves delivered to the ICU and the cost of gowns and gloves immediately prior to the start of the study.
Rate of gowns delivered to ICU per patient-day | Up to 8 months
  Number of gowns divided by patient ICU days
Rate of gloves delivered to ICU per patient-day | Up to 8 months
  Number of gloves divided by patient ICU days
Adverse events (composite of falls, medication administration errors, and pressure ulcers) | Study enrollment until study ICU discharge, truncated at 28 days after enrollment
  Composite of falls, medication administration errors, and pressure ulcers, as defined in their respective outcomes
Falls | Study enrollment until study ICU discharge, truncated at 28 days after enrollment
  Documented patient fall, regardless of degree of injury sustained
Medication administration errors | Study enrollment until study ICU discharge, truncated at 28 days after enrollment
  Documented error in administration of medications to patients, regardless of any adverse effect on the patient
Pressure ulcers | Study enrollment until study ICU discharge, truncated at 28 days after enrollment
  Documented new pressure ulcer
New MRSA colonization | Study enrollment until study ICU discharge, truncated at 28 days after enrollment
  Patient with admission surveillance culture negative for MRSA but with discharge surveillance culture positive for MRSA (collected during the final 4 months of the study).

CONTACTS AND LOCATIONS:
Overall Officials: Todd W Rice, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Huskins WC, Huckabee CM, O'Grady NP, Murray P, Kopetskie H, Zimmer L, Walker ME, Sinkowitz-Cochran RL, Jernigan JA, Samore M, Wallace D, Goldmann DA; STAR*ICU Trial Investigators. Intervention to reduce transmission of resistant bacteria in intensive care. N Engl J Med. 2011 Apr 14;364(15):1407-18. doi: 10.1056/NEJMoa1000373. PMID 21488763
- [Background] Harris AD, Pineles L, Belton B, Johnson JK, Shardell M, Loeb M, Newhouse R, Dembry L, Braun B, Perencevich EN, Hall KK, Morgan DJ; Benefits of Universal Glove and Gown (BUGG) Investigators; Shahryar SK, Price CS, Gadbaw JJ, Drees M, Kett DH, Munoz-Price LS, Jacob JT, Herwaldt LA, Sulis CA, Yokoe DS, Maragakis L, Lissauer ME, Zervos MJ, Warren DK, Carver RL, Anderson DJ, Calfee DP, Bowling JE, Safdar N. Universal glove and gown use and acquisition of antibiotic-resistant bacteria in the ICU: a randomized trial. JAMA. 2013 Oct 16;310(15):1571-80. doi: 10.1001/jama.2013.277815. PMID 24097234
- [Background] Huang SS, Septimus E, Kleinman K, Moody J, Hickok J, Avery TR, Lankiewicz J, Gombosev A, Terpstra L, Hartford F, Hayden MK, Jernigan JA, Weinstein RA, Fraser VJ, Haffenreffer K, Cui E, Kaganov RE, Lolans K, Perlin JB, Platt R; CDC Prevention Epicenters Program; AHRQ DECIDE Network and Healthcare-Associated Infections Program. Targeted versus universal decolonization to prevent ICU infection. N Engl J Med. 2013 Jun 13;368(24):2255-65. doi: 10.1056/NEJMoa1207290. Epub 2013 May 29. PMID 23718152
- [Background] Morgan DJ, Murthy R, Munoz-Price LS, Barnden M, Camins BC, Johnston BL, Rubin Z, Sullivan KV, Shane AL, Dellinger EP, Rupp ME, Bearman G. Reconsidering contact precautions for endemic methicillin-resistant Staphylococcus aureus and vancomycin-resistant Enterococcus. Infect Control Hosp Epidemiol. 2015 Oct;36(10):1163-72. doi: 10.1017/ice.2015.156. Epub 2015 Jul 3. PMID 26138329
- [Background] Derde LPG, Cooper BS, Goossens H, Malhotra-Kumar S, Willems RJL, Gniadkowski M, Hryniewicz W, Empel J, Dautzenberg MJD, Annane D, Aragao I, Chalfine A, Dumpis U, Esteves F, Giamarellou H, Muzlovic I, Nardi G, Petrikkos GL, Tomic V, Marti AT, Stammet P, Brun-Buisson C, Bonten MJM; MOSAR WP3 Study Team. Interventions to reduce colonisation and transmission of antimicrobial-resistant bacteria in intensive care units: an interrupted time series study and cluster randomised trial. Lancet Infect Dis. 2014 Jan;14(1):31-39. doi: 10.1016/S1473-3099(13)70295-0. Epub 2013 Oct 23. PMID 24161233